CLINICAL TRIAL: NCT05703503
Title: Mental Health and Healthcare in Adults With Intellectual Disabilities
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Dam Foundation (Other); University of Tromso (Other); University Hospital of North Norway (Other); The Norwegian Association for Persons with Developmental Disabilities (Unknown)
Responsible Party: Sponsor
Other Study IDs: 493747; 2022/FO387091 (Other Grant/Funding Number: Stiftelsen DAM)
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Intellectual Disabilities (F70-F79); Problem;Behaviour;Adult; Mental Health Issue; Employment; Delivery of Health Care
Keywords: Healthcare; Adults; Employment; Medication; Intellectual Disability; Neurodevelopmental Disorders
MeSH Terms: conditions — Intellectual Disability; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intellectual disability (ID) is a diagnosis characterized by significant limitations both in intellectual functioning and in adaptive behavior as expressed in conceptual, social and practical adaptive skills. The disability originates before age 18 years. The prevalence of mental ill-health among adults with intellectual disabilities is higher than the general population. Individuals with ID use psychotropic medication extensively, but studies indicate that less than one out of three who use psychotropic drugs have a psychiatric diagnosis. The drugs are usually prescribed by a regular general practitioner. People with IDs will often require health- and social services throughout their lifetimes. Studies report worse mental and physical health among people with IDs compared to the general population, in addition to more unmet healthcare needs and more difficulty accessing healthcare.

General health surveys in Norway do not include people with intellectual disabilities, and studies of health indicators in this group are largely lacking. Further, the unique organization of services for this group in Norway calls for specific research efforts. This project will use multinational health indicators for youths and adults with IDs in a biopsychosocial context in attempt to identify unmet health care needs to improve services. The project will focus on mental health and challenging behavior and how the related healthcare needs are met. We will also look at the relationship between mental health, behavioral problems and workforce employment amongst people with intellectual disabilities.

DETAILED DESCRIPTION:
Intellectual disability (ID) is a diagnosis characterized by significant limitations both in intellectual functioning and in adaptive behavior as expressed in conceptual, social and practical adaptive skills. The disability originates before age 18 years. The prevalence of mental ill-health among adults with intellectual disabilities is higher than the general population. Individuals with ID use psychotropic medication extensively, but studies indicate that less than one out of three who use psychotropic drugs have a psychiatric diagnosis. The drugs are usually prescribed by a regular general practitioner. People with IDs will often require health- and social services throughout their lifetimes. Studies report worse mental and physical health among people with IDs compared to the general population, in addition to more unmet healthcare needs and more difficulty accessing healthcare.

General health surveys in Norway do not include people with intellectual disabilities, and studies of health indicators in this group are largely lacking. Further, the unique organization of services for this group in Norway calls for specific research efforts. This project will use multinational health indicators for youths and adults with IDs in a biopsychosocial context in attempt to identify unmet health care needs to improve services. The project will focus on mental health and challenging behavior and how the related healthcare needs are met. We will also look at the relationship between mental health, behavioral problems and workforce employment amongst people with intellectual disabilities.

The following articles will be published as part of this project:

1. "The relationship between symptoms of mental health problems, diagnoses and medication in adults with intellectual disabilities"
2. "The contact between individuals with intellectual disabilities with mental health problems, and mental health professionals: characteristics of the patients and the professionals.
3. "Mental health, behavioral problems and workforce employment amongst people with intellectual disabilities".

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of intellectual disability
* Age 16 or older and providing consent to participate.

Exclusion Criteria:

* Age 15 or younger.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Persons with intellectual disabilities and registered services in the municipalities in two regions localised in the north and middle of Norway will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Health indicators in a Norwegian population of youths and adults with intellectual disabilities. | Baseline
  Health indicators as measured by The POMONA Checklist of Health Indicators (P15). The health indicators include measures of socio-demographics, Health status, Health determinants and Health systems.Physical Activity is defined as a Health determinant in this study in accordance With the POMONA Health indicator classification.

SECONDARY OUTCOMES:
The Aberrant Behaviour Checklist-Community (ABC-C) | Baseline
  The Aberrant Behaviour Checklist-Community (ABC-C) is a rating scale with 58 items for the assessment of behavioural problems in people with intellectual disabilities. The items are grouped into five subscales: (I) Irritability (15 items), (II) Social Withdrawal (16 items), (III) Stereotypic Behaviour (7 items), (IV) Hyperactivity/Non-compliance (16 items) and (V) Inappropriate Speech (4 items).
Moss Psychiatric Assessement Schedules- Checklist (MPAS- Check) | Baseline
  The checklist is a screening instrument specifically designed to help staff recognize mental health problems in the people with intellectual disability for whom they care, and to make informed referral decisions. The instrument consists of a life-events checklist and 29 symptom items scored on a four-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Erik Søndenaa, PhD, Study Chair — Department of Mental Health, Faculty of Medicine and Health Sciences, NTNU.
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway